

# TRIAL STATISTICAL ANALYSIS PLAN

c23699226-01

| BI Trial No.: | 1386-0011 |
|---|---|
| Title: | A phase I, open-label, single and multiple dose trial to investigate metabolism and pharmacokinetics of [ <sup>14</sup> C]BI 1467335 administered as oral solution in healthy male volunteers |
| | Final Protocol (Revised Protocol (based on global amendment 2)) |
| Investigational Product(s): | BI 1467335 |
| Responsible trial statistician(s): | |
| | Phone:<br>Fax: |
| | Phone:<br>Fax: |
| Date of statistical analysis plan: | 13 JUN 2018 SIGNED |
| Version: | Final |

**Proprietary confidential information** 

© 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved.

This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

TSAP for BI Trial No: 1386-0011 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| 1. | $\mathbf{T}$ | DI | $\mathbf{F} \mathbf{O}$ | FC | | TEN | TC |
|---|---|---|---|---|---|---|---|
| 1 | 1 F | ML | L O | т | $\mathbf{O}$ | | $\mathbf{I}$ |

| TITLE | PAGE | 1 |
|---|---|---|
| 1. | TABLE OF CONTENTS | 2 |
| LIST C | OF TABLES | 4 |
| 2. | LIST OF ABBREVIATIONS | |
| 3. | INTRODUCTION | |
| 4. | CHANGES IN THE PLANNED ANALYSIS OF THE STUDY | |
| <b>5.</b> | ENDPOINTS | |
| 5.1 | PRIMARY ENDPOINTS | |
| 5.2 | SECONDARY ENDPOINTS | |
| 5.2.1 | Key secondary endpoints | |
| 5.2.2 | Secondary endpoints | 9 |
| 5.3.2 | Safety parameters | 9 |
| 6.<br>6.1<br>6.2<br>6.3 | GENERAL ANALYSIS DEFINITIONSTREATMENT(S)IMPORTANT PROTOCOL VIOLATIONSSUBJECT SETS ANALYSED | 11 |
| 6.5 | POOLING OF CENTRES | 13 |
| 6.6 | HANDLING OF MISSING DATA AND OUTLIERS | |
| <b>6.7</b> | BASELINE, TIME WINDOWS AND CALCULATED VISITS | |
| <b>7.</b> | PLANNED ANALYSIS | |
| 7.1 | DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS | |
| 7.2 | CONCOMITANT DISEASES AND MEDICATION | |
| 7.3 | TREATMENT COMPLIANCE | |
| 7.4<br>7.5 | PRIMARY ENDPOINTS | |
| 7.5.1 | SECONDARY ENDPOINTS | |
| 7.5.1<br>7.5.2 | Key secondary endpoint. | |
| 7.5.2<br>7.6 | Secondary endpoints | |
| 7.6.1 | | |
| 7.0.1<br>7.7 | Safety endpointsEXTENT OF EXPOSURE | |
| 7.7<br>7.8 | SAFETY ANALYSIS | |
| 7.8.1 | Adverse events | |
| 7.8.2 | Laboratory data | |
| 7.8.2<br>7.8.3 | Vital signs | |
| 7.8.4 | ECG | |
| 7.8.5 | Others | |
| 1.0.3 | Our 5 | IJ |

# Boehringer Ingelheim TSAP for BI Trial No: 1386-0011

| | P for BI Trial No: 1386-0011 | |
|---|---|---|
| Proprieta | ary confidential information © 2018 Boehringe | r Ingelheim International GmbH or one or more of its affiliated companies |
| 8. | REFERENCES | 20 |
| | | 21 |
| 10. | HISTORY TABLE | 22 |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1386-0011 
Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# LIST OF TABLES

| Table 6.1: 1 | Flow chart of analysis phases for statistical analyses of AEs, safety | |
|---|---|---|
| | laboratory data and vital signs | 11 |
| Table 6.2: 1 | Important protocol violations | 12 |
| Table 6.3: 1 | Subject sets analysed | 13 |
| Table 10: 1 | History table | 22 |

TSAP for BI Trial No: 1386-0011 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### LIST OF ABBREVIATIONS 2.

| Term | Definition / description |
|---|---|
| ADPC | Proper name of the analysis dataset containing PK concentrations per time-point or per time-interval |
| ADPP | Proper name of the analysis dataset containing calculated PK parameters |
| ADS | Analysis dataset |
| AE | Adverse Event |
| AESI | Adverse event of special interest |
| $\mathrm{AUC}_{0	ext{-}	au}$ | area under the concentration-time curve of the analyte over the time interval from $\boldsymbol{\tau}$ |
| AUC0-tz | Area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point |
| BI | Boehringer Ingelheim |
| BLQ | Below the lower limit of quantification |
| BRPM | Blinded Report Planning Meeting |
| CARE | Clinical data analysis and reporting environment |
| Cmax | Maximum measured concentration of the analyte in plasma |
| $C_{\text{max,ss}}$ | maximum measured concentration of the analyte at steady state |
| CRF | Case Report Form |
| CTP | Clinical Trial Protocol |
| CTR | Clinical Trial Report |
| CV | Arithmetic coefficient of variation |
| ECG | Electrocardiogram |
| fe <sub>faeces</sub> , 0-t2 | fraction of [ <sup>14</sup> C]-radioactivity excreted in faeces as percentage of the administered oral dose over the time interval from 0 to the last quantifiable time point |
| fe <sub>urine, 0-t2</sub> | fraction of [14C]-radioactivity excreted in urine as percentage of the administered oral dose over the time interval from 0 to the last quantifiable time point |
| gCV | Geometric coefficient of variation |
| gMean | Geometric mean |
| ICH | International Conference On Harmonisation |
| MedDRA | Medical Dictionary For Regulatory Activities |
| NOA | Not analysed |

TSAP for BI Trial No: 1386-0011 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

| Term | Definition / description |
|-------|----------------------------------------|
| NOR | No valid result |
| NOS | No sample available |
| PK | Pharmacokinetics |
| PKS | Pharmacokinetic parameter analysis set |
| PSTAT | Project Statistician |
| PT | Preferred Term |
| PV | Protocol Violation |
| Q1 | Lower Quartile |
| Q3 | Upper Quartile |
| RAGe | Report appendix generator |
| SD | Standard Deviation |
| SDL | Subject data listing |
| SOC | System Organ Class |
| TS | Treated Set |
| TSAP | Trial Statistical Analysis Plan |
| ULN | Upper limit of normal range |

TSAP for BI Trial No: 1386-0011

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 3. INTRODUCTION

As per ICH E9 (1), the purpose of this document is to provide a more technical and detailed elaboration of the principal features of the analysis described in the revised CTP, and to include detailed procedures for executing the statistical analysis of the primary and secondary variables and other data.

This TSAP assumes familiarity with the CTP and its amendments. In particular, the TSAP is based on the planned analysis specification as written in CTP Section 7 "Statistical Methods and Determination of Sample Size". Therefore, TSAP readers may consult the CTP for more background information on the study, e.g., on study objectives, study design and population, treatments, definition of measurements and variables, planning of sample size, randomisation.

CRF data entered by the site will be stored in a trial database within the Oracle Clinical<sup>TM</sup> system. Electronically transferred data will be stored in CDR.

The statistical analyses will be performed within the validated working environment CARE, including SAS<sup>TM</sup> (current Version 9.4, by SAS Institute Inc., Cary, NC, USA), and a number of SAS<sup>TM</sup>-based tools (e.g., macros for the analyses of AE data or laboratory data; Report Appendix Generator system (RAGe) for compilation/formatting of the CTR appendices).

PK parameters will be calculated using Phoenix WinNonlin<sup>TM</sup> software (version 6.3, Certara USA Inc., Princeton, NJ, USA).

#### 4. CHANGES IN THE PLANNED ANALYSIS OF THE STUDY

All analyses described in this TSAP are in accordance with the statistical methods described in the revised CTP.

#### 5. ENDPOINTS

#### 5.1 PRIMARY ENDPOINTS

Primary endpoints are PK endpoints as defined in Section 5.5.1.1 of the CTP:

- $fe_{urine, 0-t2}$  (fraction of  $[^{14}C]$ -radioactivity excreted in urine as percentage of the administered oral dose over the time interval from 0 to the last quantifiable time point)
- $fe_{faeces, 0-12}$  (fraction of [ $^{14}$ C]-radioactivity excreted in faeces as percentage of the administered oral dose over the time interval from 0 to the last quantifiable time point)

**CTP**: Timeframe: The timeframe for determination of these endpoints depends on discharge of radioactivity from each individual subject and is predicted to vary between 2-7 weeks after drug administration.

#### 5.2 SECONDARY ENDPOINTS

#### 5.2.1 Key secondary endpoints

Not applicable.

#### 5.2.2 Secondary endpoints

Secondary PK endpoints will be defined as in Section 5.5.1.2 of the CTP.

Secondary endpoints in the single dose treatment group are  $C_{max}$  and  $AUC_{0-tz}$  of total radioactivity and  $C_{max}$  and  $AUC_{0-tz}$  of BI 1467335 in plasma.

Secondary endpoints in the multiple doses treatment group are  $C_{max}$  and  $AUC_{0-tz}$  of total radioactivity and  $C_{max.ss}$  and  $AUC_{0-\tau}$  of BI 1467335 in plasma.

#### 5.3.2 Safety parameters

Further safety parameters of interest will be used as defined in Section 5.2.1 of the CTP:

#### CTP:

- AEs (including clinically relevant findings from the physical examination)
- Safety laboratory tests
- 12-lead ECG
- *Vital signs (blood pressure, pulse rate)*

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1386-0011 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

TSAP for BI Trial No: 1386-0011

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 6. GENERAL ANALYSIS DEFINITIONS

#### 6.1 TREATMENT(S)

For basic study information on treatments to be administered, assignment of treatment groups, and selection of doses, cf. Section 4 of the CTP.

Subjects were planned to be treated either with

- a single dose of [<sup>14</sup>C]BI 1467335 (10 mg BI 1467335 calculated as free base) or
- multiple dose of 10 mg BI 1467335 and a single dose of [<sup>14</sup>C] BI 1467335 (10 mg BI 1467335 calculated as free base) on Day 28

Subjects in the multiple doses treatment group will receive unlabelled 10 mg BI 1467335 as film-coated tablet once daily from Day 1 to Day 27. In the morning of Day 28, following an overnight fast of at least 10 h, the subjects will receive one single oral dose of the radiolabelled trial drug. Treatment with nonradiolabelled compound (film-coated tablets) will continue from Day 29 up to Day 40, but may be stopped earlier in case release criteria have been met, cf. Section 3.1 of the CTP.

For statistical analysis of AEs, safety laboratory data and vital signs, the following analysis phases are defined for each subject:

Table 6.1: 1 Flow chart of analysis phases for statistical analyses of AEs, safety laboratory data and vital signs

| Study analysis phase | Label | Start (inclusive) | End (exclusive) |
|---|---|---|---|
| Screening | Screening | Date of informed consent | Date/time of administration of study drug |
| On-treatment | 10 mg BI SD, or<br>10 mg BI MD,<br>respectively | Date/time of administration of study drug | 0:00 AM on day after subject's trial termination date |

Appendix 16.1.13.1.8.1 and Appendix 16.1.13.1.8.2 AE displays will present results for the on-treatment phase only. CTR Section 15 will present results for the screening and on-treatment phase.

In CTR Section 15 AE tables (but not in Appendix 16.1.13.1.8.1 and Appendix 16.1.13.1.8.2 AE tables), the following total will be provided in addition:

- "Total on-trt BI", defined as the total over all on-treatment phases involving BI 1467335
- "Total", defined as the total over all study phases (incl. screening and on-treatment).

More details on the technical implementation of these analyses are provided in the ADS Plan of this TSAP.

#### 6.2 IMPORTANT PROTOCOL VIOLATIONS

Consistency check listings (for identification of violations of time windows) and a list of protocol deviations (e.g. deviations in drug administration) will be provided to be discussed at the RPM/DBLM. At this meeting, each protocol deviation must be assessed to determine whether it is an IPV. For definition of IPVs, and for the process of identification of these, refer to the BI reference document "Protocol Violation Handling Definitions" (2).

Table 6.2: 1 Important protocol violations

| Cat<br>/ Co | egory | Description |
|---|---|---|
| | ouc | |
| A | | Entrance criteria not met |
| | A1 | Inclusion criteria violated |
| | A2 | Exclusion criteria violated |
| B | | Informed consent |
| | B1 | Informed consent not available |
| | B2 | Informed consent too late |
| C Trial medication and randomisation | | Trial medication and randomisation |
| | C1 | Incorrect trial medication taken |
| | C3 | Non-compliance |
| | C4 | Incorrect intake of trial medication |
| D | | Concomitant medication |
| | D1 | Prohibited medication use |
| E | | Missing data |
| | | None <sup>1</sup> |
| G | | Other trial specific important violations |
| | G1 | Certain violations of procedures used to measure secondary PK data |

Violations C1, C2 and G1 can only be detected at the trial site.

Source: BI reference document "Protocol Violation Handling Definitions" (2).

If any IPVs are identified, they are to be summarised into categories and will be captured in the RPM/DBLM minutes via an accompanying Excel spreadsheet (3). The table above contains the categories which are considered to be IPVs in this trial. If the data show other IPVs, this table will be supplemented accordingly by the time of the RPM/DBLM.

IPVs will be summarised and listed.

<sup>&</sup>lt;sup>1</sup> Missing visits, evaluations, and tests will be considered missing data, not PVs

#### 6.3 SUBJECT SETS ANALYSED

All entered subjects who received study medication will be included in the safety analysis and in the PK analysis depending on the availability of measurement values, and on their adherence to the CTP.

The following subject sets will be defined for statistical analysis:

#### • Treated set (TS):

This subject set includes all subjects who received at least one dose of study drug. This is the full analysis set population in the sense of ICH-E9. It will be used for analysis of safety, demographic data and baseline characteristics.

## • Pharmacokinetic parameter set (PKS):

This subject set includes all subjects in the TS who provide at least one primary or secondary PK parameter that was not excluded because of PVs relevant to the statistical evaluation of PK endpoints as defined in Section 7.3 of the CTP.

The discussion of all exceptional cases and problems and the decisions on the allocation of subjects to analysis sets will be made at latest at the RPM/DBLM.

Table 6.3: 1 Subject sets analysed

| | Subj | ect set |
|---------------------------------|------|---------|
| Class of endpoint | TS | PKS |
| Disposition | X | |
| Exposure | X | |
| IPVs | X | |
| Demographic/baseline endpoints | X | |
| Primary and secondary endpoints | | X |
| Safety parameters | X | |

#### 6.5 POOLING OF CENTRES

This section is not applicable, because the study was performed in only one centre.

#### 6.6 HANDLING OF MISSING DATA AND OUTLIERS

**CTP**: If a subject is removed from or withdraws from the trial prior to first administration of trial medication, the data of this subject will not be entered in the case report form (CRF) or

trial database and will not be reported in the clinical trial report (CTR). If a subject is removed from or withdraws from the trial after first administration of trial medication, this will be documented and the reason for discontinuation must be recorded in the CRF. In this case, the data will be included in the CRF/trial database and will be reported in the CTR.

**CTP**: With respect to safety evaluations, it is not planned to impute missing values.

The only exceptions where imputation might be necessary for safety evaluation are AE dates. Missing or incomplete AE dates are imputed according to BI standards (4).

Missing data and outliers of PK data are handled according to BI standards (5).

#### Plasma / Urine concentration-time tables

**CTP**: Drug concentration data identified with NOS (no sample available), NOR (no valid result), NOA (not analysed), or BLQ (below the lower limit of quantification) will be displayed as such and not replaced by zero at any time point (this rule also applies also to the lag phase, including the predose values).

#### Pharmacokinetic parameters

**CTP**: Drug concentration data identified with NOS, NOR or NOA will generally not be considered. Concentration values in the lag phase identified as BLQ will be set to zero. All other BLQ values of the profile will be ignored. The lag phase is defined as the period between time zero and the first time point with a concentration above the quantification limit.

#### 6.7 BASELINE, TIME WINDOWS AND CALCULATED VISITS

For safety measurements baseline is defined as the last measurement before first study drug administration.

Time windows are defined in Section 6.1 of the CTP. Adherence to time windows will be checked at the RPM/DBLM.

#### 7. PLANNED ANALYSIS

The format of the listings and tables will follow the BI guideline "Reporting of clinical trials and project summaries"  $(\underline{6})$ .

The individual values of all subjects will be listed. Listings will generally be sorted by dose group, subject number and visit (if visit is applicable in the respective listing). AE listings will be sorted by assigned treatment (see <u>Section 7.8.1</u> below for details). The listings will be contained in Appendix 16.2 (SDL) of the CTR.

The following standard descriptive statistical parameters will be displayed in summary tables of continuous variables:

N number of non-missing observations

Mean arithmetic mean SD standard deviation

Min minimum Median median Max maximum

For plasma concentrations as well as for all PK parameters the following descriptive statistics will additionally be calculated:

CV arithmetic coefficient of variation

gMean geometric mean

gCV geometric coefficient of variation

The data format for descriptive statistics of plasma concentrations will be identical with the data format of the respective concentrations. The descriptive statistics of PK parameters will be calculated using the individual values with the number of decimal places as provided by the evaluation program. Then the individual values as well as the descriptive statistics will be reported with three significant digits in the CTR.

Tabulations of frequencies for categorical data will include all possible categories and will display the number of observations in a category as well as the percentage (%) relative to the respective treatment group. Percentages will be rounded to one decimal place. The category missing will be displayed if and only if there actually are missing values. Percentages will be based on all subjects in the respective subject set whether they have non-missing values or not.

#### 7.1 DEMOGRAPHIC AND OTHER BASELINE CHARACTERISTICS

Only descriptive statistics are planned for this section of the CTR. These will be based on the TS.

#### 7.2 CONCOMITANT DISEASES AND MEDICATION

Concomitant diseases will be coded according to the most recent version of MedDRA. Concomitant medication will be coded according to the most recent version of the World Health Organisation – Drug Dictionary.

Only descriptive statistics are planned for this section of the CTR.

A medication will be considered concomitant to a treatment, if it

- is ongoing at the time of administration of the respective treatment or
- starts within the analysis phase of the respective treatment (see <u>Section 6.1</u> for a definition of treatments and analysis phases).

#### 7.3 TREATMENT COMPLIANCE

Treatment compliance will not be analysed as a specific endpoint. Any deviations from complete intake will be addressed in the RPM/DBLM (cf. <u>Section 6.2</u>) and described in the CTR.

#### 7.4 PRIMARY ENDPOINTS

Only descriptive statistics are planned for this section of the CTR. These will be based on the PKS. The analysis of standard PK parameters is performed according to BI standards (5) [001-MCS-36-472 RD-01].

#### Exclusion of PK parameters

The ADS ADPP contains column variables APEXC and APEXCO indicating inclusion/exclusion (APEXC) of a PK parameter and an analysis flag comment (APEXCO). All analyses based on the PKS are based on PK parameter values which are not flagged for exclusion, i.e. with APEXC equal to "Included".

#### Exclusion of plasma concentrations

The ADS ADPC (PK concentrations per time-point or per time-interval) contains column variables ACEXC or ACEXCO indicating inclusion/exclusion (ACEXC) of a concentration and an analysis flag comment (ACEXCO). Exclusion of a concentration depends on the analysis flag comment ACEXCO. For example, if ACEXCO is set to "ALL CALC", the value will be excluded for all types of analyses based on concentrations. If ACEXCO is set to "DESC STATS" the value will be excluded from descriptive evaluations per planned time point/time interval. If ACEXCO contains the addition "TIME VIOLATION" or "TIME DEVIATION", the value can be used for further analyses based on actual times. If ACEXCO is set to "HALF LIFE", the value will be excluded from half-life calculation only; the value is included for all other analyses. Excluded concentration itself will be listed in the CTR associated with an appropriate flag.

Further details are given in "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies" (5) and "Description of Analytical Transfer Files and PK/PD Data Files" (7).

#### 7.5 SECONDARY ENDPOINTS

#### 7.5.1 Key secondary endpoint

Not applicable.

#### 7.5.2 Secondary endpoints

Only descriptive statistics are planned for this section of the CTR. These will be based on the PKS.

#### 7.6 FURTHER ENDPOINTS

#### 7.6.1 Safety endpoints

Further safety endpoints will be analysed as described in Section 7.8 of this TSAP.

#### 7.7 EXTENT OF EXPOSURE

Only descriptive statistics are planned for this section of the CTR.

#### 7.8 SAFETY ANALYSIS

All safety analyses will be performed on the TS.

#### 7.8.1 Adverse events

AEs will be coded with the most recent version of MedDRA.

The analyses of AEs will be descriptive in nature. All analyses of AEs will be based on the number of subjects with AEs and not on the number of AEs.

For analysis, multiple AE occurrence data on the eCRF will be collapsed into one event provided that all of the following applies:

- All AE attributes are identical (lower level term, intensity, action taken, therapy required, seriousness, reason for seriousness, relationship, outcome, AESI)
- The occurrences were time-overlapping or time-adjacent (time-adjacency of two occurrences is given if the second occurrence started at most 1 hour after the first occurrence ended)

For further details on summarization of AE data, please refer to "Analysis and Presentation of Adverse Event Data from Clinical Trial" (8) [001-MCG-156] and "Handling of missing and incomplete AE dates" (4) [001-MCG-156 RD-01].

The analysis of AEs will be based on the concept of treatment emergent AEs. That means that all AEs will be assigned to the screening phase or on-treatment phase as defined in Section 6.1.

An overall summary of AEs will be presented. This overall summary will comprise summary statistics for the class of other significant AEs according to ICH E3 and for the class of AESIs.

**CTP:** The following are considered as AESIs in this trial:

Hepatic injury

A hepatic injury is defined by the following alterations of hepatic laboratory parameters:

- o an elevation of AST and/or ALT  $\geq$ 3-fold ULN combined with an elevation of total bilirubin  $\geq$ 2-fold ULN measured in the same blood sample, and/or
- $\circ$  aminotransferase (ALT, and/or AST) elevations  $\geq$ 10 fold ULN.

The investigator had to classify on the eCRF whether an observed AE was an AESI or not.

According to ICH E3 (9), AEs classified as "other significant" need to be reported and will include those non-serious and non-significant AEs

- (i) which are marked haematological or other lab abnormalities, or
- (ii) which were reported with "action taken = discontinuation" or "action taken = reduced", or
- (iii) which lead to significant concomitant therapy as identified by the Clinical Monitor/Investigator at a Medical Quality Review Meeting.

The frequency of subjects with AEs will be summarised by treatment, primary SOC and preferred term. AEs which were considered by the investigator to be drug related will be summarised separately. Separate tables will also be provided for subjects with SAEs, subjects with AESIs and subjects with other significant AEs (according to ICH E3 (9)). The frequency of subjects with AEs and the frequency of subjects with AEs considered by the investigator to be drug related will also be summarised by maximum CTCAE grade, primary SOC and preferred term.

The SOCs and preferred terms within SOCs will be sorted by descending frequency overall treatment groups.

For disclosure of AE data on ClinicalTrials.gov, the frequency of subjects with non-serious AEs occurring with an incidence of greater than 5 % (in preferred terms) will be summarised by treatment, primary SOC and preferred term. The frequency of subjects with SAEs will also be summarised.

For disclosure of AE data in the EudraCT register, the frequency of AEs, the frequency of non-serious AEs with an incidence of greater than 5 % (in preferred terms) and the frequency of SAEs will be summarised.

#### 7.8.2 Laboratory data

The analyses of laboratory data will be descriptive in nature and will be based on BI standards "Display and Analysis of Laboratory Data" (10).

Analyses will be based on normalised values, which means transforming to a standard unit and a standard reference range.

Descriptive statistics of laboratory values over time and for the difference from baseline (see <u>Section 6.7</u>) will be provided. Frequency tables of changes between baseline and the value two weeks after last study drug intake (i.e., Day 15 for SD group and Day 43 for MD group) with respect to the reference range will be presented.

Possibly clinically significant abnormal laboratory values are only those identified either in the Investigator's comments or at the RPM/DBLM at the latest. It is the Investigator's responsibility to decide whether a lab value is clinically significant abnormal or not. Standard or project-specific rules for flagging clinically significant values in an automated manner will not be applied in this study.

Clinically relevant findings in laboratory data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

### 7.8.3 Vital signs

The analyses of vital signs (blood pressure and pulse rate) will be descriptive in nature. Descriptive statistics of vital signs over time and for the difference from baseline (see Section 6.7) will be provided.

Clinically relevant findings in vital signs data will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

#### 7.8.4 ECG

Abnormal findings in ECG will be reported as baseline conditions (at screening) or as AEs (during the trial) if judged clinically relevant by the investigator, and will be analysed as such.

#### **7.8.5** Others

Physical examination findings will be reported as relevant medical history/baseline condition (i.e., a condition already existent before intake of study drug) or as AE and will be summarised as such. No separate listing or analysis of physical examination findings will be prepared.

TSAP for BI Trial No: 1386-0011 

Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 8. **REFERENCES**

| 1 | CPMP/ICH/363/96: "Statistical Principles for Clinical Trials", ICH Guideline Topic E9, Note For Guidance on Statistical Principles for Clinical Trials, current version. |
|---|---|
| 2 | 001-MCS-50-413_RD-01: "Protocol Violation Handling Definitions", current version; IDEA for CON |
| 3 | 001-MCS-50-413_RD-02: "Important Manual Protocol Violations Spreadsheet", current version; IDEA for CON |
| 4 | 001-MCG-156_RD-01: "Handling of missing and incomplete AE dates", current version; IDEA for CON. |
| 5 | 001-MCS-36-472_RD-01: "Noncompartmental Pharmacokinetic / Pharmacodynamic Analyses of Clinical Studies", current version; IDEA for CON |
| 6 | 001-MCG-159: "Reporting of Clinical Trials and Project Summaries", current version; IDEA for CON |
| 7 | 001-MCS-36-472_RD-03: "Description of Analytical Transfer Files and PK/PD Data Files", current version; IDEA for CON |
| 8 | 001-MCG-156: "Analysis and Presentation of Adverse Event Data from Clinical Trial", current version; IDEA for CON |
| 9 | CPMP/ICH/137/95: "Structure and Content of Clinical Study Reports", ICH Guideline Topic E3; Note For Guidance on Structure and Content of Clinical Study Reports, current version |
| 10 | 001-MCG-157: "Handling, Display and Analysis of Laboratory Data", current version; IDEA for CON. |

# **Boehringer Ingelheim**

TSAP for BI Trial No: 1386-0011 
Proprietary confidential information © 2018 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### HISTORY TABLE **10.**

Table 10: 1 History table

| Version | Date<br>(DD-MMM-YY) | Author | Sections changed | Brief description of change |
|---|---|---|---|---|
| Final | 13-JUN-18 | | None | This is the final TSAP without any modification |